CLINICAL TRIAL: NCT04299867
Title: Perioperative Tissue Penetration of Antimicrobials in Infants
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00103890
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Bowel Dysfunction
MeSH Terms: conditions — Intestinal Diseases | interventions — Metronidazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples Intestinal tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- < 34 weeks gestational age: Metronidazole will be given per standard of care prior to incision. Intraoperative plasma samples will be obtained from pre-existing vascular access catheters at end of bolus, 30, 60, 90 minutes, at time of intestinal excision(s), and at the end of the case in ethylenediaminetetraacetic acid microcontainers, exceeding no more than approximately 5 mL total.
  At the time of intestinal excision, the surgeon will cut at least 500 mg of intestine from the specimen, ensuring all layers of bowel are included. If more than one intestinal sample is taken during the surgery, such as in the case of multiple strictures removed, each sample will be obtained and labeled appropriately.
  Interventions: Procedure: Bowel Surgery with Metronidazole
- 34 weeks gestational age: Metronidazole will be given per standard of care prior to incision. Intraoperative plasma samples will be obtained from pre-existing vascular access catheters at end of bolus, 30, 60, 90 minutes, at time of intestinal excision(s), and at the end of the case in ethylenediaminetetraacetic acid microcontainers, exceeding no more than approximately 5 mL total.
  At the time of intestinal excision, the surgeon will cut at least 500 mg of intestine from the specimen, ensuring all layers of bowel are included. If more than one intestinal sample is taken during the surgery, such as in the case of multiple strictures removed, each sample will be obtained and labeled appropriately.
  Interventions: Procedure: Bowel Surgery with Metronidazole

INTERVENTIONS:
Procedure: Bowel Surgery with Metronidazole — Metronidazole will be given per standard of care prior to incision. Intraoperative plasma samples will be obtained from pre-existing vascular access catheters at end of bolus, 30, 60, 90 minutes, at time of intestinal excision(s), and at the end of the case in ethylenediaminetetraacetic acid microcontainers, exceeding no more than approximately 5 mL total.
  At the time of intestinal excision, the surgeon will cut at least 500 mg of intestine from the specimen, ensuring all layers of bowel are included. If more than one intestinal sample is taken during the surgery, such as in the case of multiple strictures removed, each sample will be obtained and labeled appropriately.

SUMMARY:
This study aims to define the pharmacokinetic (PK) properties of a commonly used antibiotic to treat cIAI, metronidazole, in the intestinal wall tissue of healthy infants undergoing intestinal surgery to optimize intestinal wall penetration of antibiotics in infants. Metronidazole will be given at standard of care intravenous loading dose of 30 mg/kg 15 minutes prior to incision, with a maximum dose of 2g. Intraoperative plasma samples will be obtained from pre-existing vascular access catheters at end of bolus, 30, 60, 90 minutes, at time of intestinal excision, and at the end of the case in ethylenediaminetetraacetic acid microcontainers, exceeding no more than 5mL total.

DETAILED DESCRIPTION:
This is a single center pilot pharmacokinetic (PK) study to concomitantly measure antibiotic concentrations in the plasma and the intestinal wall of healthy infants undergoing intestinal surgery.

Metronidazole will be given at standard of care intravenous loading dose of 30 mg/kg 15 minutes prior to incision, with a maximum dose of 2g. Exact time, dose, and infusion rate and duration will be recorded. The use of a loading dose will allow characterization of plasma and tissue PK after a single dose that would be expected with steady state dosing, thus increasing the translatability of the investigator's findings to cIAI treatment.

Intraoperative plasma samples will be obtained from pre-existing vascular access catheters at end of bolus, 30, 60, 90 minutes, at time of intestinal excision, and at the end of the case in ethylenediaminetetraacetic acid microcontainers, exceeding no more than 5mL total. At the time of intestinal excision, the surgeon will cut at least 250mg of intestine from the specimen, ensuring all layers of bowel are included. This sample will be placed in a sterile, dry container. All samples will be processed and stored in a -80°C freezer within 1 hour of acquisition. Samples will be batched and shipped to a central commercial laboratory (OpAns Analytical Solutions LLC, Durham, NC) for concentration measurement of metronidazole and its primary metabolite 2-hydroxymetronidazole using a HPLC/MS/MS plasma assay previously developed and validated per FDA guidance. This assay will be modified and validated for tissue concentration measurement utilizing porcine intestinal tissue and run over three mediums to ensure correct measurement. The samples will also be used to quantify CYP2A6 protein levels using commercially available enzyme-linked immunosorbent assay kits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0 to 2 years at enrollment
2. Written informed consent provided by a parent or legal guardian
3. Scheduled to undergo elective intestinal operation for the removal of non-infected bowel
4. Sufficient intravascular access to complete the study procedures

Exclusion Criteria:

1. Prior treatment with metronidazole for any dose during the 72 hours prior to study drug administration.
2. Patients with active inflammatory or infectious conditions of the bowel such as inflammatory bowel disease, Hirschprung's disease in the portion of bowel to be excised, diverticular disease, cancerous or pre-cancerous lesions, colitis, enteritis, ulcerative disease, Meckel's diverticulum, celiac disease, and irritable bowel syndrome.
3. Renal dysfunction defined as serum creatinine >2 mg/dL at enrollment
4. Receiving any extracorporeal life support including extracorporeal membrane oxygenation, ventricular assist devices, and renal replacement therapy at enrollment
5. Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the data.

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children < 2 years of age undergoing intestinal surgery
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Clearance | Day of Surgery + 12 hours
Pharmacokinetic Half-life | Day of Surgery + 12 hours
Pharmacokinetic Volume of Distribution | Day of Surgery + 12 hours
Pharmacokinetic Area under the curve | Day of Surgery + 12 hours

SECONDARY OUTCOMES:
CYP2A6 quantification | Day of Surgery + 12 hours
Ratio of Metronidazole to 2-hydroxymetronidazole concentration | Day of Surgery + 3-4 hours
Mean Plasma Concentration of Metronidazole | Day of Surgery + 3-4 hours
Mean Plasma Concentration of 2-hydroxymetronidazole | Day of Surgery + 3-4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hornik, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data and results will be shared in publication

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT04299867/Prot_SAP_ICF_000.pdf